CLINICAL TRIAL: NCT04520087
Title: Evaluation of Clinical and Radiographic Results After Surgical Treatment With Implant-free Allograft for Anterior Shoulder Dislocation: Pilot Study
Brief Title: Clinical and Radiographic Assessment After Surgical Treatment of Anterior Shoulder Dislocation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J-Plasty
Record Dates: First submitted 2020-07-29; First posted 2020-08-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Anterior Shoulder Dislocation; Bone Defects; Shoulder Instability
Keywords: Implant-Free Shoulder Instability; Bone Grafting; Shoulder Instability; Glenoid; allograft
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allograft fixation (Experimental): Patients with anteroinferior shoulder instability will be clinically treated with a mini-open arthrotomic technique involving the fixation of the corticospongeous bone graft on the glena.
  Interventions: Procedure: allograft fixation

INTERVENTIONS:
Procedure: allograft fixation — Patients with anteroinferior shoulder instability will be clinically treated with a mini-open arthrotomic technique involving the fixation of the corticospongeous bone graft on the glena.
  Other Names: bone grafting for shoulder instability

SUMMARY:
The purpose of this study is to evaluate the clinical and radiographic results after surgical treatment with implant-free allograft in the treatment of Anterior Shoulder Dislocation and to assess the safety of the surgery.

DETAILED DESCRIPTION:
Patients will be informed about the study and potential risks. All patients giving written informed consent will undergo a screening visit to assess the eligibility criteria.

Patients who meet the eligibility requirements will perform a pre-treatment visit in order to assess their healthy state. Also, patients will undergo to the radiographic visit (RX and TX) as request by clinical practice.

All the patients will be treated with arthrotomy mini-open technique with bone allograft at the site of the shoulder lesion.

After surgery all the patients will be followed up to 24 months through clinical and radiographic visits.

ELIGIBILITY:
Inclusion Criteria:

* antero.inferior shoulder instability with bone loss

Exclusion Criteria:

* Patients incapable of understanding or wanting;
* Patients suffering from: rheumatic diseases, diabetes, infectious processes, congenital ligament laxity, epilepsy, severe osteoporosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in DASH score at 24th months | 24 months
  The Disabilities of the Arm, Shoulder and Hand (DASH) Score is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.

SECONDARY OUTCOMES:
Change from baseline in DASH score | Baseline, 1, 3, 6, and 12 months
  The Disabilities of the Arm, Shoulder and Hand (DASH) Score is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Change from Baseline in Constant score | Baseline, 1, 3, 6, 12 and 24 months
  The Constant score contains both physician-completed and patient-reported portions. The four domains include pain (15 possible points), activities of daily living (20 possible points), mobility (40 possible points), and strength (25 possible points). Scores range from 0 points (most disability) to 100 points (least disability).
Change from Baseline in Rowe score | Baseline, 1, 3, 6, 12 and 24 months
  The Rowe score is a 3-item physician completed instrument. Its questions address the categories of shoulder stability, motion, and function. Scores range from 0 to 100 with a score of 90-100 points indicating an excellent evaluation, 75-89 points indicating a good evaluation, 51-74 points indicating a fair evaluation, and 0-50 points indicating a poor evaluation.
Change from Baseline in EQ-5D-3L (EuroQoL) CurrentHealthAssessment: | Baseline, 1, 3, 6, 12 and 24 months
  EQ-5D is a standardized instrument for measuring generic health status. The classification system defines health in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each dimension with three levels ("no problems" [level 1], "some problems" [level 2], and "extreme problems" [level 3]), resulting in a total of 243 (3^5) health states. The 3L classification system defined the 243 health states by combining different levels from each dimension, with 11111 and 33333 representing full health and worst health, respectively.
Evaluation of the grade of the Shoulder Osteoarthritis through Kellgren-Lawrence scoring | 24 months
  The Kellgren and Lawrence system is a common method of classifying the severity of osteoarthritis (OA).
  The K-L system defines OA in 5 grades:
  grade 0 (none): definite absence of x-ray changes of osteoarthritis grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping grade 2 (minimal): definite osteophytes and possible joint space narrowing grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends grade 4 (severe): large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends.
Evaluation of the Allograft integration | 6 and 12 months
  Radiographic signs of allograft integration through the CT-dual energy instrument at 6 and 24 month post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Guerra, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy